University Hospitals of Leicester

Leicester Royal Infirmary Infirmary Square Leicester LE1 5WW

## **Consent Form**

IRAS Project ID: 256620

Study Number:

taking consent

| Participant Identification Number | er: | | |
|---|---|---|---|
| Study Title: The efficacy of cream in alleviating the pain of | | ctrical Nerve Stimulation ver<br>njections in adults - A Randon | |
| Principle Investigator: Ms Rajshree Jayarajan Plo | | | Please initial the boxes |
| 1. I confirm that I have read and Version 2.0 (v2.0) for the above information, ask questions and h | study. I have had the | opportunity to consider the | |
| 2. I understand that my particip time without giving any reason, | _ | | |
| 3. I understand that relevant second looked at by responsible individuals or from regulatory authorities we permission for these individuals | uals from the study to | eam, the sponsor, NHS Trust, my taking part in the research. | I give |
| 4. I wish to receive details of the | results of the study a | and agree to be contacted | |
| by letter or email | Yes No | | |
| 5. I agree to take part in the above | e study | | |
| Name of Participant | Date | Signature | |
| Name of Researcher | <br>Date | Signature | <u>—</u> |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes
Informed Consent Form V2.0 17/02/2019 Transcutaneous Electrical Nerve Stimulation for Local Anaesthetic TENS-LA

University Hospitals of Leicester Wiss

Leicester Royal Infirmary Infirmary Square Leicester LE1 5WW